CLINICAL TRIAL: NCT06280248
Title: Study of Different Modalities of Endoscopic Ultrasound (EUS)-Guided Post-pancreatitis Pancreatic Fluid Collection Drainage
Brief Title: EUS Guided Drainage of Post Pancreatitis Pancreatic Fluid Collection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Abodief, Assiut university Hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUS in pancreatic fluid
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pancreas Pseudocyst
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic ultrasound guided cystogastrostomy of symptomatic pancreatic pseudocyst (Other)
  Interventions: Procedure: Endoscopic ultrasound guided cystogastrostomy of symptomatic pancreatic pseudocyst

INTERVENTIONS:
Procedure: Endoscopic ultrasound guided cystogastrostomy of symptomatic pancreatic pseudocyst — The technical success rates, clinical success rates, and potential complications of the different endoscopic ultrasound-guided techniques for the best drainage of pancreatic fluid collections (PFCs) as regard type, caliber, and number of plastic stents and the ideal timing for stent removal will be assessed.
  Also compare early vs. late intervention for complete endoscopic necrosectomy of walled off pancreatic necrosis (WOPN ) as regard to technical success rates, clinical success rates, potential complications, and the number of sessions needed will be done.
  In order to evaluate total resolution or a reduction in cyst diameters with clinically significant improvement in symptoms, patients will be monitored for one month and six months following the insertion of the stent.

SUMMARY:
The number as well as the caliber of plastic stents used for EUS-guided PFC drainage are controversial in current practice [Lin et al., 2014]. The timing of necrosectomy in WOPN drainage continues to be debated. To date, no comparative studies have been conducted to investigate the ideal timing for stent removal. Thus, the aim of our study is to:

* Assess the technical success rates, clinical success rates and potential complications of the different techniques for the best drainage of PFCs as regard type, caliber and number of plastic stents and ideal timing for stent removal.
* Compare between early vs late intervention for complete endoscopic necrosectomy of WOPN as regard technical success rates, clinical success rates, potential complications and number of sessions needed.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) accounts for over 50% of all hospital admissions for pancreatic disease and still represents one of the most unpredictable diseases of the digestive system (NICE guideline, 2018). Therefore, AP can be linked to a number of systemic or local problems; in its most severe form, it can result in multiple organ failure and even death (Rana et al., 2015).

Pancreatic fluid collections (PFCs) are a common complication of AP, with a reported incidence of 43% (Cui et al., 2014). When there is pancreatic damage, such as AP, pancreatic trauma, postsurgery, posttransplant, or occlusion of the pancreatic duct (PD), PFCs develop. The management of PFCs must be guided by the classification of these entities according to their acuity and the presence or absence of necrosis.

Surgical drainage has been the standard of care for PFCs. The paradigm has, however, changed in favor of methods requiring endoscopic intervention and minimally invasive drainage due to recent advancements in endoscopic tools and techniques (Cui et al., 2014).

The Atlanta criteria refer to the initial global agreement on PFC classification that was created in 1993. PFCs were categorized as acute (forming within 4 weeks of pancreatitis onset) or chronic (forming after 4 weeks of pancreatitis onset) based on the original Atlanta criteria. Pancreatic necrosis, pancreatic pseudocysts (PPs), or pancreatic abscesses were the three further subtypes of chronic PFCs (Bradley et al., 1993).

Recent advances in pathophysiology and diagnostic tools warranted a revision to these criteria. The most important distinction to arise from the new classification system, known as the revised Atlanta criteria (Banks et al., 2013), is the delineation between collections containing only fluid and collections containing necrotic tissue with or without accompanying fluid.

The criteria for acute versus chronic PFCs is preserved, but new additions have been made based on the presence of necrosis. Acute collections are divided into acute peripancreatic fluid collections and acute necrotic collections. Chronic collections are divided into PPs and walled-off pancreatic necroses (WOPNs). These distinctions have helped guide the development of treatment strategies tailored to the acuity and contents of a given collection (Banks et al., 2013).

The original Atlanta criteria recommended drainage for PFCs based on the size of the collection as well as the presence of symptoms including abdominal pain, gastrointestinal (GI) or biliary obstruction, vascular compression, or infection. With recent advances in diagnostic tools and interventional techniques, indications for the drainage of PFCs have been revised to emphasize the presence of symptoms or infected collection (Trikudanathan et al., 2019).

1) Symptomatic sterile collections with or without the presence of necrosis; symptoms include persistent abdominal pain, ileus, and gastric outlet obstruction with or without fever.

(2) Proven or suspected infected PFCs with or without the presence of necrosis. Asymptomatic sterile necrotic collections and asymptomatic WOPN are not recommended for drainage, as they may undergo spontaneous resolution given time (Freeman et al., 2012).

The reason is that among asymptomatic necrosis, the content is liquefied in 28-35% of cases and the size decreases, especially in extra-pancreatic WON or WON without a disconnected pancreatic duct, without the need for further necrosectomy (Pawar et al., 2021).

According to a recent meta-analysis (Nakai et al., 2023), early interventions (before 4 weeks) for necrotizing pancreatitis were associated with higher mortality, the same rate of adverse events, and clinical success compared to delayed interventions; however, another meta-analysis reported similar outcomes for early or delayed interventions but a longer hospital stay for early interventions (Ramai et al., 2023).

As EUS can precisely quantify the distance between the GI lumen and the pseudocyst and use Doppler US to define a safe nonvascular window for draining, it is the recommended method for evaluating PFCs (Giovannini et al., 2007). Similarly, the type of stent that is selected for drainage can also be directly impacted by the sort of fluid that EUS detects.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic sterile PFCs; symptoms include persistent abdominal pain, ileus, and gastric outlet obstruction with or without fever.
* Proven or suspected infected PFCs with or without the presence of necrosis.
* Patients with pancreatic pseudocyst that unresolved for at least 6 weeks after the last episode of pancreatitis and making compression on surrounding organs such as common bile duct (CBD), portal vein (PV).

Exclusion Criteria:

* Patient refusal.
* Patients with major comorbidities being unfit for general anesthesia.
* Patients with moderate to marked ascites.
* Patients with bleeding tendencies and impaired coagulation profile.
* Patients with proven or suspected malignant pancreatic neoplasms.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Complete resolution or a decrease in the sizes of pancreatic fluid collections (PFCs) | 2 year
  * Achievement of complete resolution or a decrease in the sizes of pancreatic fluid collections (PFCs) with clinical symptomatic improvement after 1 month and 6 months of stent placement using different EUS PFCs drainage techniques.
  * Compare the technical and clinical success rates and potential complications of the different techniques of EUS guided pancreatic fluid collections (PFCs) drainage.